CLINICAL TRIAL: NCT00821392
Title: A Randomized, Multi-Center, Double Blinded, Allopurinol-Controlled, Placebo-Controlled Parallel Group, 5-Arm, Dose-Response,Bridging Study to Assess the Efficacy and Safety of Febuxostat in Subject With Gout
Brief Title: Phase III Trial of Febuxostat in Korea Gout Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SK Chemicals Co., Ltd. (Industry)
Responsible Party: SK Chemicals Co.,Ltd., SK Chemicals Co.,Ltd.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TMX-67
Record Dates: First submitted 2009-01-12; First posted 2009-01-13 (Estimated); Last update posted 2009-01-13 (Estimated); Status verified 2007-10

CONDITIONS: Gout
MeSH Terms: conditions — Gout | interventions — Febuxostat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (5):
- 1 Febuxostat 40mg (Active Comparator)
  Interventions: Drug: Febuxostat
- 2 Febuxostat 80mg (Active Comparator)
  Interventions: Drug: Febuxostat
- 3 Febuxostat 120mg (Active Comparator)
  Interventions: Drug: Febuxostat
- 4 Allopurinol 300mg (Sham Comparator)
  Interventions: Drug: Febuxostat
- 5 Placebo (Placebo Comparator)
  Interventions: Drug: Febuxostat

INTERVENTIONS:
Drug: Febuxostat

SUMMARY:
This study was designed to evalute the efficacy and safety of Febuxostat after oral administration to patientd with gout in Korea

DETAILED DESCRIPTION:
This is a multi-center, randomized, double-blind, allopurinol and placebo controlled, parallel, 5 arms, dose response, bridging study of 4 weeks duration.

If subjects pass the screening evaluation after submitting a signed informed consent, they will be randomly assigned to one of the five treatment regimens; febuxostat 40mg, 80mg, 120mg, placebo or allopurinol 300mg. Colchicine 0.6mg QDis given to minimize the risk of gout flares during the washout/run-in period and during the double study period.

ELIGIBILITY:
Inclusion Criteria:

<Day -14>

1. age :18-85 years
2. female: either post-menopausal for at least 2 years, surgically sterile, or using a medically accepted means of contraception
3. female: negative serum pregnancy test
4. subjects who satisfy ARA (American Rheumatism Association)
5. subjects must have a renal function defined as: serum creatinine ≤ 1.5 mg/dL <Day -1>

1.serum urate level ≥8.0mg/dL 2.creatinine level ≤ 1.5mg/dL 3.subject continued to meet all inclusion and no exclusion criteria

Exclusion Criteria:

1. women who are breast-feeding or pregnant
2. a history of xanthinuria
3. allopurinol intolerance
4. receiving thiazide diuretic therapy
5. secondary hyperuricemia
6. required > 10mg/day of prednisone during the study stable dose(≤10mg/day), inhaled and intranasal steroids will be allowed.
7. concomitant therapy containing aspirin or other salicylates(systemic or topical, prescribed or non-prescribed) stable, low doses aspirin will be allowed(i.e. ≤325mg/day).
8. any change in hormone replacement therapy or oral contraceptive therapy within 3 months of the screening visit
9. alcohol intake≥ 14drinks/week alcohol abuse within 5 years or current excessive alcohol use was prohibited.
10. concomitant therapy with any urate-lowering therapy
11. active liver disease or hepatic dysfunction : ALT, AST ≥1.5 ULN
12. subject was unable to take colchicine or contradictory to colchicine
13. a serum urate level < 8.0mg/dL and not taking uric acid lowering therapy
14. rheumatoid arthritis or any active arthritis requiring for the medication treatment
15. a history of cancer (other than basal cell carcinoma of the skin) within 5 years prior to the screening visit, or had taken any systemic cancer chemotherapy within 5 years prior to the screening visit
16. participated in another investigational trial within the 30days prior to the screening visit
17. any other significant medical condition as defined by the investigator

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2006-08; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)